CLINICAL TRIAL: NCT05806957
Title: Pivotal Trial to Assess the Clinical Performance of Ophthal-360
Brief Title: Pivotal Trial to Assess the Clinical Performance of Ophthal-360 for the Detection of Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ophthalytics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CD0001
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Fluorescein Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Device: Color Fundus Photography with Non-Mydriatic and Mydriatic Cameras
  Interventions: Device: Fundus Photography

INTERVENTIONS:
Device: Fundus Photography — Subjects will undergo Fundus Photography using FDA approved non-mydriatic fundus cameras and mydriatic camera with OCT

SUMMARY:
Multicenter, prospective, study to assess the performance of the Ophthal-360 platform in the diagnosis of more-than-mild Diabetic Retinopathy (mtmDR) in diabetic patients with no previous diagnosis of DR.

DETAILED DESCRIPTION:
This is a multicenter, prospective study in which 500 adult subjects at risk for DR but never before diagnosed who satisfy all entry criteria will be enrolled at up to 5 primary care sites.

An additional sub-study will be performed on 30 subjects to assess the precision of the algorithm in detecting DR by imaging these subjects multiple times to demonstrate intra- and inter-operator reliability of the algorithm.

All enrolled subjects will undergo retinal imaging by a novice operator with no experience using the fundus cameras listed. Images from each retinal imaging device will be saved to a computer and uploaded to the server for evaluation by the Ophthal-360 service. A report will be generated and archived for the results of each image.

After imaging by the novice operator, each patient will then have their eyes photographed by a professional fundus photographer using standard mydriatic and OCT imaging for macular edema evaluation. These images will be sent to a Fundus Photography Reading Center for final determination and diagnosis. Patients will received the result of the FPRC evaluation, but not be provided the reports generated by the software.

A comparison between the FPRC determination and the software generated report will be performed to evaluate the analytical performance of the algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 22 years old.
2. A documented history of Diabetes Mellitus, defined as any of the following:

   * Hemoglobin A1c (HbA1c) ≥ 6.5% based on repeated assessments
   * Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L) based on repeated assessments
   * Oral Glucose Tolerance test with 2-hour plasma glucose ≥ 200 mg/dL (11.1mmol/L) using equivalent of 75g anhydrous glucose dose in water.
   * Symptoms of hyperglycemia or hyperglycemic crisis with random plasma glucose ≥ 200mg/dL (11.1 mmol/L)
   * Criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA).
3. Willing to undergo fundus photography by up to 4 different methods and/or cameras.
4. Has signed a written informed consent form prior to study participation.

Exclusion Criteria:

1. Diagnosed with uncorrectable vision loss (e.g., with the use of eyeglasses), blurred vision, or floaters.
2. Diagnosed with macular edema, severe non-proliferative retinopathy, proliferative retinopathy, radiation retinopathy, or retinal vein occlusion.
3. Has a positive history for laser treatment of the retina or injections into either eye, or any history of retinal surgery.
4. Is currently participating in another investigational eye study and actively receiving investigational product for DR or Diabetic Macular Edema (DME).
5. Has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia or previous enucleation).
6. Is contraindicated for imaging by fundus imaging systems used in the study:

   * hypersensitive to light
   * recently (within 6 months) underwent photodynamic therapy (PDT)
   * taking medication that causes photosensitivity
   * positive history for angle-closure glaucoma or narrow anterior chamber angles

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with diabetes at risk for diabetic retinopathy but not previously diagnosed.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the Ophthal-360 Software to detect diabetic retinopathy in fundus images | 1 day
  Performance of the Ophthal-360 Software when compared to results of evaluation of fundus photographs by qualified experts.
Specificity of the Ophthal-360 Software to detect diabetic retinopathy in fundus images | 1 day
  Performance of the Ophthal-360 Software when compared to ground truth evaluation of fundus photographs by qualified experts.

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared.